CLINICAL TRIAL: NCT01113515
Title: An Interventional, Placebo-Controlled, Randomized, Double-blinded Dose Comparison, Phase I/II Study to Determine the Safety and Efficacy of a New Gel Formulation of Esmolol Hydrochloride (Galnobax®) for the Treatment of Diabetic Foot Ulcer (DFU)
Brief Title: Clinical Investigation of Galnobax® for the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novalead Pharma Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Novalead-Galnobax-0210
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer; Diabetic wound; chronic non healing ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo gel
- Galnobax 20% QD (Experimental): Esmolol Hydrochloride (Galnobax) 20% gel once daily
  Interventions: Drug: Esmolol hydrochloride
- Galnobax 20% BID (Experimental): Esmolol Hydrochloride (Galnobax) 20% gel twice daily
  Interventions: Drug: Esmolol hydrochloride
- Galnobax 14% BID (Experimental): Esmolol Hydrochloride (Galnobax) 14% gel twice daily
  Interventions: Drug: Esmolol hydrochloride

INTERVENTIONS:
Drug: Esmolol hydrochloride
  Other Names: Galnobax-14%
  Arms: Galnobax 14% BID
Drug: Esmolol hydrochloride
  Other Names: Galnobax-20%
  Arms: Galnobax 20% BID
Drug: Esmolol hydrochloride
  Other Names: Galnobax-QD
  Arms: Galnobax 20% QD
Drug: Placebo gel
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine safety and efficacy of a new gel formulation of Esmolol hydrochloride (Galnobax®) for the treatment of Diabetic Foot Ulcer (DFU). The study will compare number and types of adverse events occured, rates of wound closure and percentage of wounds closed in Galnobax treated groups versus placebo group.

DETAILED DESCRIPTION:
This is an interventional, placebo-controlled, randomized, double-blinded, dose comparison, phase I/II study of Galnobax® in subjects with diabetic foot ulcers. Additionally the effect of dosage and frequency of application will also be studied . The total trial duration per subject is 25 weeks which comprises of 1 week for screening, 12 weeks of treatment and 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 95 years, inclusive, with Type 1 or Type 2 diabetes undergoing therapy for glycemic control
* Subjects having below knee ulcer of at least 4 week and maximum of 52 weeks duration which is a full thickness ulcer without exposure of bone, muscle, ligaments, or tendons
* Ulcer should be clinically non-infected
* Ulcer area (length x width) measurement between 1.5 cm2 and 10 cm2, inclusive and post debridement ulcer area less than or equal to 12 cm2.
* Full-thickness ulcer of Grade 1 or Grade 2 as per Wagner's classification system
* Recently debrided ulcer (2 weeks prior to screening) and post debridement ulcer free of necrotic debris, foreign bodies, sinus tracts, tunneling, and undermining, comprised of healthy vascularized tissue as determined by the Investigator
* Inability to perceive 10 grams pressure using Semmes-Weinstein 5.07 monofilament in the peri-ulcer area
* Ankle Brachial index between 0.7 and 1.2

Exclusion Criteria:

* Actively infected ulcers with or without purulent discharge, ulcers with exposed bone or associated with osteomyelitis.
* Subjects having cellulitis, ischemic or gangrenous ulcers in the opinion of the Investigator
* Glycosylated hemoglobin (HbA1C) >12%
* Diagnosed and/ currently unstable hypotension, heart block, cardiac failure, and other cardiac complications
* Subject diagnosed with cancer undergoing chemotherapy
* Revascularization surgery 4 weeks prior to signing the ICF
* Renal failure as defined by serum creatinine >3.0 mg/dL or renal insufficiency requiring frequent dialysis
* Poor nutritional status as measured by serum albumin <3.0 g/dL
* Active Charcot or other structural deformity that would prevent adequate off-loading of the study foot

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2015-06-27 (Actual); Study Completion 2015-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vickie R Driver, DPM FACFAS, Principal Investigator — Providence Veteran Affairs Medical Center, RI
Locations (5):
- VA New England Health Care Division, Providence, Rhode Island, United States
- India (3):
  - S.L. Raheja Hospital, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Center, Pune, Maharashtra
  - M V Hospital for Diabetes Pvt. Ltd., Chennai, Tamil Nadu
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Rastogi A, Kulkarni SA, Deshpande SK, Driver V, Barman H, Bal A, Deshmukh M, Nair H. Novel Topical Esmolol Hydrochloride (Galnobax) for Diabetic Foot Wound: Phase 1/2, Multicenter, Randomized, Double-Blind, Vehicle-Controlled Parallel-Group Study. Adv Wound Care (New Rochelle). 2023 Aug;12(8):429-439. doi: 10.1089/wound.2022.0093. Epub 2022 Nov 16. PMID 36245145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID
Started | 10 | 9 | 14 | 11
Completed | 10 | 9 | 10 | 10
Not Completed | 0 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID | Total
Number analyzed (Participants) | 10 | 9 | 14 | 11 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (9.37) | 50.0 (5.85) | 56.2 (11.56) | 53.0 (7.75) | 53.5 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 9
  Male | 8 | 7 | 12 | 8 | 35
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 1 | 1 | 2
  Malaysia | 1 | 1 | 2 | 1 | 5
  India | 9 | 8 | 11 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome
Description: Number of participant with adverse events (AEs) till end of follow-up phase in different groups
Time Frame: Till end of follow up period (Week 25)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID
Number analyzed (Participants) | 10 | 9 | 14 | 11
Participants | 1 | 3 | 9 | 6

2. Secondary Outcome: Efficacy Outcome
Description: To evaluate the percent change in ulcer area and ulcer volume from baseline till end of treatment (Week 12) in different groups
Time Frame: Baseline and end of treatment (Week 12 or 84 +/- 2 days)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID
Number analyzed (Participants) | 10 | 9 | 10 | 10
percent change
  Percent Change in Ulcer Area | 80.67 (34.09) | 82.58 (31.57) | 95.80 (9.85) | 86.56 (35.07)
  Percent Change in Ulcer Volume | 84.57 (32.99) | 55.41 (92.31) | 83.36 (39.60) | 99.40 (1.70)

3. Secondary Outcome: Efficacy Outcome
Description: Time in days taken for closure of wound in different groups from baseline till end of treatment (week 12 or 84 +/- 2 days)
Time Frame: From baseline till end of treatment (Week 12 or 84 +/- 2 days)
Measure: Median (Full Range); unit: days
Groups:
- Galnobax 20% QD: Esmolol Hydrochloride (Galnobax) 20% gel once daily
  Esmolol hydrochloride
- Galnobax 20% BID: Esmolol Hydrochloride (Galnobax) 20% gel twice daily
  Esmolol hydrochloride
- Galnobax 14% BID: Esmolol Hydrochloride (Galnobax) 14% gel twice daily
  Esmolol hydrochloride
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID
Number analyzed (Participants) | 6 | 5 | 5 | 6
days | 53.5 [22 to 72] | 77 [8 to 86] | 72 [23 to 84] | 49.5 [29 to 85]

4. Other Pre Specified Outcome: Pharmacokinetic Measurements
Description: Pharmacokinetic profile of Galnobax® in subset of patients suffering from DFU
Time Frame: pre-dose (prior to first study drug application), and at 15 and 30 minutes, 1, 3, 6, 12, and 24 hours after the first study drug application on day 0, weeks 1, 4, and 12 (prior to study drug application).
Measure: Mean (Standard Deviation); unit: Cmax (ng/mL) of Esmolol acid
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID
Number analyzed (Participants) | 4 | 4 | 4 | 4
Cmax (ng/mL) of Esmolol acid | 0.0 (0.0) | 78.451 (83.176) | 113.802 (117.383) | 340.018 (430.944)

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | Placebo | Galnobax 20% QD | Galnobax 20% BID | Galnobax 14% BID
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 4/14 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 3/9 | 6/14 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Galnobax 20% QD (N=9) | Galnobax 20% BID (N=14) | Galnobax 14% BID (N=11)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Galnobax 20% QD (N=9) | Galnobax 20% BID (N=14) | Galnobax 14% BID (N=11)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceradaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has prepared an integrated clinical/statistical report. As this was a multicenter study, any publication/presentation of data was to include the entire study population. Publication/presentation of data from individual study centers is not allowed without explicit permission from the sponsor.